CLINICAL TRIAL: NCT05732584
Title: Effect of Auditory Stimulation by Family Voices in Preventing Delirium Among Sedative Patients in Emergency Intensive Care Units ：A Randomized Controlled Trial
Brief Title: Effect of Auditory Stimulation by Family Voices in Preventing Delirium: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-1013
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Delirium
Keywords: Delirium; Intensive Care Units; Auditory Stimulation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- structured family voice stimulation (Experimental): Patients in this group were provided with structured family voice stimulation
  Interventions: Other: structured family voice stimulation
- unstructured family voice stimulation (Experimental): Patients in this group were provided with unstructured family voice stimulation
  Interventions: Other: unstructured family voice stimulation
- Control group (No Intervention): Patients in this group will receive no specific voice stimulation

INTERVENTIONS:
Other: structured family voice stimulation — The structured family voice stimulation is played to the patients for the first five days after admission to eicu until transfer out or death. The content of the recording is developed according to the structured script.
  Arms: structured family voice stimulation
Other: unstructured family voice stimulation — The unstructured family voice stimulation is played to the patients for the first five days after admission to eicu until transfer out or death.
  Arms: unstructured family voice stimulation

SUMMARY:
Delirium is an acute cerebral dysfunction syndrome characterized by acute fluctuating changes in consciousness, cognitive dysfunction, and disorientation. It's especially common in critically ill patients of emergency intensive care units and seriously threatens the survival and prognosis of patients and causes heavy economic burdens to the family, society, and medical service system. Impaired verbal communication, unfamiliar medical personnel, physical restraint, spatial-temporal disorientation, mechanical ventilation and sedation medication use can lead to a lack of adequate sensory stimulation and a high risk of delirium. Acoustic stimulation as a non-invasive non-pharmacological intervention can provide some sensory stimulation as a surrogate for critically ill patients. This research designs the content scripts from the needs of ICU patients and families for sound stimulation. The goal of this randomized controlled study is to test the effect of auditory stimulation by family voices in preventing delirium among sedative patients in emergency Intensive care units.

DETAILED DESCRIPTION:
Patients are separated from their families and society under the closed management of the intensive care unit, the use of sedative drugs, mechanical ventilation, impaired verbal communication, physical restraint, environmental noise, and prolonged light exposure, which lead to a lack of adequate sensory stimulation, causing sensory deprivation in patients to some extent. In turn, sensory deprivation may cause multisensory perceptual confusion and hallucinations, affecting patients' orientation and thinking and triggering delirium, so providing appropriate sensory stimulation to critically ill patients may help to improve patients' orientation and attention, correct patients' thinking confusion and prevent delirium, and in clinical practice, sensory stimulation is considered as an important part of multicomponent delirium prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* transferred to the EICU from emergency admission
* no other history of emergency, surgery, or ICU admission history within 30 days
* no delirium in the first screening of Emergency Intensive Care Unit(EICU) admission
* with an expected length of stay in EICU longer than 24h and use of sedation medication

Exclusion Criteria

* Presence of hearing impairment, severe dementia, psychiatric disorder, or other severe brain dysfunction that hinders delirium assessment
* persistent coma or deep sedation (RASS score of -4 to -5)
* patients without a family member who can cooperate with the recording
* external ear disease or surgery that hinders earphone wearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
incidence of delirium | up to 5 days
  use the Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
delirium severity | up to 5 days
  use Confusion Assessment Method for the Intensive Care Unit 7-item (CAM-ICU-7), ranging from 0-7 , higher scores means higher delirium severity.
delirium duration | up to 5 days
  use the Confusion Assessment Method for the ICU (CAM-ICU)
delirium-free days | up to 5 days
  use the Confusion Assessment Method for the ICU (CAM-ICU)
delirium subtype | up to 5 days
  use the Confusion Assessment Method for the ICU (CAM-ICU) and Richmond Agitation Sedation Scale(RASS)
time to first delirium | up to 5 days
  use the Confusion Assessment Method for the ICU (CAM-ICU)
family anxiety levels | up to 5 days
  families were assessed using the Self-Rating Anxiety Scale (SAS) at the beginning and at the end of the intervention. (The score ranges from 25 to 100 and higher scores means more anxious situation)
family depression levels | up to 5 days
  families were assessed using the Self-Rating Depression Scale (SDS) at the beginning and at the end of the intervention. (The score ranges from 25 to 100 and higher scores means more depressed situation)
Duration of mechanical ventilation | up to 5 days
  Duration of use of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jingfen Jin, Master, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No